CLINICAL TRIAL: NCT07199153
Title: Accuracy of 3D Printed Custom-Made Registration Method for Dynamic Navigation Implant Surgery Using Mininavident in the Esthetic Zone: A Clinical Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sherif Aly Sadek (Other)
Collaborators: Cairo University (Other)
Responsible Party: Sponsor-Investigator, Sherif Aly Sadek, Associate Professor, Cairo University
Organization: Cairo University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-4-24
Record Dates: First submitted 2025-09-13; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Dental Implantation Accuracy
Keywords: Dynamic Navigation Surgery; Dental Implant Surgery; Implant Accuracy; Esthetic Zone; Computer-Guided Implantology; Digital Dentistry; Prosthetically Driven Implant Planning

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 3D Printed Registration for Dynamic Navigation Surgery (Experimental): Participants with a single missing anterior maxillary tooth will undergo implant placement using the Mininavident dynamic navigation system with a custom-made, 3D printed registration marker. The marker enables registration of CBCT and intraoral scans for prosthetically driven implant planning and real-time guided surgery.
  Interventions: Device: D Printed Custom Registration Marker for Dynamic Navigation

INTERVENTIONS:
Device: D Printed Custom Registration Marker for Dynamic Navigation — A patient-specific, 3D printed registration marker designed for use with the Mininavident dynamic navigation system. The marker is fabricated based on CBCT and intraoral scans, enabling accurate registration between virtual planning and clinical implant placement in the esthetic zone. Accuracy of placement is assessed through postoperative CBCT superimposition.

SUMMARY:
This clinical trial evaluates the accuracy of a 3D printed custom-made registration method for dynamic navigation implant surgery using the Mininavident system in the esthetic zone of the anterior maxilla. Ten patients with a single missing anterior tooth will undergo CBCT-based planning, intraoral scanning, and guided implant placement using 3D printed registration markers. Postoperative CBCT analysis will measure deviations between planned and placed implants in terms of angular, coronal, and apical positions. The study aims to determine whether 3D printed markers provide clinically acceptable accuracy (<2 mm, <5°) and to assess their feasibility as a reproducible alternative to standard registration methods.

DETAILED DESCRIPTION:
Accurate implant positioning is essential for esthetic and functional success, particularly in the anterior maxilla. Dynamic navigation systems (DNS) provide real-time guidance but depend on reliable registration between patient anatomy and virtual planning. Errors may occur with conventional fiducial markers, highlighting the need for more precise methods.

This clinical trial investigates the use of 3D printed custom registration markers with the Mininavident DNS for implant placement in the esthetic zone. Ten patients with a single missing anterior tooth will undergo CBCT-based planning and guided implant placement using the custom markers. Postoperative CBCT scans will be compared with preoperative plans to measure positional and angular deviations.

The primary outcome is the accuracy of implant placement, with deviations expected to remain within clinically acceptable limits (<2 mm, <5°). Secondary outcomes include assessing the feasibility and reproducibility of incorporating 3D printed registration into DNS workflows. Results may validate this approach as a cost-effective, patient-specific solution to enhance precision and predictability in implant dentistry.

ELIGIBILITY:
Inclusion Criteria:

* Single missing tooth in the anterior maxilla
* ≥12 mm bone height and ≥5.5 mm width
* D3 bone density
* Angle's Class I occlusion
* No systemic contraindications to implant surgery

Exclusion Criteria:

* Heavy smoking or uncontrolled diabetes
* Radiation therapy involving the head and neck
* Parafunctional habits (e.g., bruxism)
* Class III malocclusion or edge-to-edge bites

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-08-10 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-10-15 (Estimated)

PRIMARY OUTCOMES:
Accuracy of Implant Placement Using 3D Printed Registration Markers | Within 1 week after implant placement
  Accuracy will be assessed by measuring deviations between the planned and actual implant positions using postoperative CBCT superimposed with the preoperative plan.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Only de-identified, aggregate data (summary of implant deviation measurements and feasibility outcomes) will be shared. No individual participant-level raw data will be made available. Data may be provided upon reasonable request to the principal investigator for academic or scientific purposes